CLINICAL TRIAL: NCT06095557
Title: Discovery Study of Using a Magnetocardiography (MCG) Device at Emergency Departments (EDs)
Brief Title: MCG Discovery Study in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SB Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SB-ACS-002
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: ACS - Acute Coronary Syndrome; NSTEMI - Non-ST Segment Elevation MI
Keywords: magnetocardiography; MCG
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sponsor MCG device (Experimental): All participants will receive a scan from the Sponsor MCG device
  Interventions: Device: Sponsor MCG device

INTERVENTIONS:
Device: Sponsor MCG device — unshielded device measuring cardiac magnetic fields

SUMMARY:
This prospective discovery study is designed to demonstrate the feasibility of using an unshielded, mobile MCG device in an Emergency Department (ED) setting. The main question it aims to answer is whether interpretable data can be reliably collected as part of an ED workflow.

ELIGIBILITY:
Inclusion Criteria:

* Presents to ED with symptoms of Acute Coronary Syndrome (ACS)
* Can provide written consent

Exclusion Criteria:

* Presents to ED with ST-Elevation Myocardial Infarction (STEMI)
* Presents to ED with Atrial Fibrillation
* Clear non-ischemic cause for symptoms (i.e. trauma)
* Active thoracic metal implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
% analyzable Sandbox MCG data | during the procedure (MCG scan)
  % Sandbox MCG data collected and suitable for analysis

SECONDARY OUTCOMES:
Sandbox MCG safety | 30 days
  Device-related adverse events
Characterization of scan results that may differentiate between high risk and low risk ACS patients | during the procedure (MCG scan)
  Signal Noise Ratio of ECG features
Characterization of scan results that may differentiate between high risk and low risk ACS patients | during the procedure (MCG scan)
  t-wave field maximum angle
Characterization of scan results that may differentiate between high risk and low risk ACS patients | during the procedure (MCG scan)
  heartbeats needed to obtain signal

CONTACTS AND LOCATIONS:
Overall Officials: Kit Yee Au-Yeung, PhD, Study Director — SB Technology, Inc.
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No